CLINICAL TRIAL: NCT02448134
Title: A Community-Based Strategy for Preventing Underage Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AA021726 (NIH)
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Youth Access (Experimental): Youth Engagement in Prosocial Alcohol-Free Activities Participate in the "Reward and Reminder" program in their community
  Interventions: Behavioral: Youth Access
- Control (No Intervention): Student will receive regular information and programs.

INTERVENTIONS:
Behavioral: Youth Access — Community youth will participate in various school-and-community-wide pro-social, anti-alcohol activities.
  Arms: Youth Access

SUMMARY:
This project evaluates a combination of policy and social influence interventions to reduce adolescent alcohol use and its sequelae.

DETAILED DESCRIPTION:
1. In this community-wide intervention, we will evaluate a comprehensive underage alcohol use reduction intervention that combines policy and enforcement elements focused on 1) reducing social and commercial access to alcohol, and 2) increasing the likelihood of legal sanctions associated with use and misuse, and 3) mobilize parental and peer influences not to use. We will work with 6 communities in Lane County. Schools in the 6 communities will be randomly assigned to receive the intervention immediately, or to be part of a wait list control group. If the results of the intervention are promising, we will partner with Lane County Prevention to bring the intervention to the wait list schools after 2 years.

   Our project aims to encourage the participation of youth in a number of different activities that will be conducted, for the most part, outside of school hours. These activities will help youth to discover, on their own, some of the risks and issues related to excessive alcohol use. Teams of youth will interview community members (e.g., law enforcement, health care workers, business leaders, etc.) about some of the problems that can accompany excessive alcohol use. The youth will present their results to the City Council, School Board, the student body, etc., and attempt to build support for more aggressive city ordinances against underage drinking (e.g., increased penalties for serving to minors) and for stepped-up enforcement of existing laws (e.g., drunk driving). Youth will also interview parents regarding their beliefs and expectations related to alcohol use, and will advocate for alcohol-free social events organized by the school or community members. Teams will post updates on their progress on social media, increasing awareness among the student body, and will compete for various awards and prizes. In prior work done in school districts throughout Oregon over the past twenty-five years, we have found that these strategies are effective in preventing youth use of tobacco, alcohol, and other drugs.

   This project has several key elements:

   Community and Youth Engagement in Prosocial Alcohol-Free Activities Project staff will work with school and community representatives to help organize diverse teams of youth volunteers who will lead activities related to (a) learning about and increasing awareness about the dangers of alcohol use, (b) pushing for policy change and enforcement with the goal of reducing alcohol access, use and consumption (e.g., tougher laws for DUII) and (c) creating fun, alcohol-free recreational opportunities for all youth . Youth volunteers will be actively consented to participate teams. We will work with existing community coalitions, where possible, to promote sustainability. We will use social media to spread the news about the progress of the youth teams and activities. A project-monitored Facebook page will be part of each community's effort to communicate about recreation activities, reward prosocial youth behavior, and promote safer norms and behavior around alcohol use. Further description of Team Activities is attached.

   Reducing Access to Alcohol in the Community Project staff will work with local law enforcement and youth to focus on the enforcement of laws and the promotion of norms that can reduce the problems of alcohol misuse in the community. ORI will work with Lane County Prevention to conduct purchase surveys in which young-looking 21-year olds attempt to purchase alcohol, and track whether or not clerks are willing to sell at various outlets in the recruited communities. In intervention communities, youth teams may be involved in soliciting local businesses to provide rewards for clerks who obey the law and do not sell. This "Reward and Reminder" program has been successfully used to reduce illegal sales of tobacco and alcohol to minors in communities in Oregon and Wyoming. Lane County is currently preparing to test the use of Reward and Reminder in reducing illegal alcohol, tobacco and lottery sales. In control communities, we will conduct purchase surveys. Surveys will take place once a year.

   Current Youth Alcohol Use and Proximal Measures Bi-monthly student surveys of Alcohol Access and Attitudes: Students in 9th - 11th grade will complete a 20-minute survey on alcohol use and intentions to use, perceived access to alcohol, perceptions of the dangers of alcohol misuse, and perceptions of peer, parent and community attitudes about youth misuse of alcohol, every two months for two years. (See attached proposed measure). Student data will be tracked over time. Parents will be mailed a letter in advance to provide information about the project, and they will have an option to have their child opt out of the survey.

   Baseline and follow up anonymous data on youth alcohol use will be obtained from the state of Oregon from the Oregon Student Wellness Survey and the OSAS survey (formerly Oregon Healthy Teens Survey). These two anonymous statewide surveys alternate each year, but items related to alcohol use and attitudes are asked in both surveys. We will work with the Oregon Department of Education and the superintendents of schools in each community to have access to this secondary data source. The survey is taken in 6th, 8th and 11th grades all over the state of Oregon. We will use both 8th and 11th grade survey data to get a snapshot of current alcohol use and intentions to use in our communities (8th grade data from spring of 2014 is a baseline for 9th graders in the 2014-2015 school year). The data is anonymous and will give us a good snapshot of current use and intentions to use.
2. Describe the research hypothesis (es) or the specific aims(s). The specific aims of the project are to: a) experimentally evaluate a comprehensive strategy to reduce underage drinking and alcohol-related problems in 6 communities; b) assess the effects of the intervention on intermediate outcomes that represent proximal outcomes of the interventions, such as sales to minors, perceived alcohol availability, perceive community norms, alcohol expectancies, and perceptions of the social attractiveness non-drinking teens; and c) analyze the extent to which intermediate outcomes mediate the observed effects of the prevention strategies on alcohol use and problems.
3. Describe the relevance of the research to previous and/or continuing work in the field. This proposal aligns with the movement to integrate policy-oriented interventions with programs targeting individual psychological functioning. Evidence shows that fully implementing policies to increase the costs of obtaining and using alcohol (e.g., penalty for use, difficulty obtaining) has preventive effects, although some of that may result from changes in the normative beliefs and attitudes of people. Ample evidence indicates that substance use can be deterred by increasing the degree to which parents communicate expectations and set limits and by school-based programs targeting social influences and relevant attitudes. It is thus natural to develop and test interventions that marshal as many of the known influences on the problem as we can. Considering that these intervention effects, though empirically established, are modest, it is vital to explore whether combining them can produce additive effects resulting in a greater impact on adolescent alcohol use than these types of interventions can produce on their own. At the same time, we need efficient strategies that can be maintained. This project will combine a policy-focused intervention with an innovative and efficient strategy to mobilize peer and parental influences to not drink. The policy component is designed to reduce youth access to alcohol and increase the perceived likelihood of sanctions via intensified enforcement and rewards for compliance with underage drinking laws.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be enrolled in 9th through 11th grade in the 6 recruited communities. In year 02, we will add entering 9th graders at the same schools, and will follow 11th graders into 12th grade. We will also make use of secondary data for 8th and 11th graders.

Exclusion Criteria:

* None

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7379 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in frequency (days per month; drinks per day) of underage alcohol use | Bi-Annually, over two years
  Alcohol Access and Attitudes Survey
  Youth indicated their alcohol use over the previous 30 days (i.e., "In the last 30 days, on how many days have you consumed alcoholic beverages?"). Response options included none, zero times (0), occasionally, maybe one to three times (1), fairly often, about four to six times (2), regularly, seven to nine times (3), and all the time, ten or more times (4).

SECONDARY OUTCOMES:
Change in attitudes regarding acceptability of underage alcohol use | Bi-Annually, over two years
  Alcohol Access and Attitudes Survey
Reward and Reminder: Value of Law Enforcement in Preventing Youth Alcohol Use | Bi-Annually, over two years
  Alcohol sales outlets were assessed by confederates in terms of their willingness to sell alcohol to young-looking individuals who did not possess a valid ID (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Biglan, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States